CLINICAL TRIAL: NCT04379128
Title: Attentional Impairment in People With Epilepsy
Acronym: ETAPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02748-49
Record Dates: First submitted 2020-04-27; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with epilepsy: Attentional tasks : D2-R task and TAP battery (sustained attention, alertness, divided attention) executive task : digit span, incompatibility and flexibility task (TAP battery), verbal fluencies depression score (NDDI-E scale) and anxiety score (GAD-7 scale)
  Interventions: Other: Attentional tasks
- Normal controls: Attentional tasks : D2-R task and TAP battery (sustained attention, alertness, divided attention) executive task : digit span, incompatibility and flexibility task (TAP battery), verbal fluencies depression score (NDDI-E scale) and anxiety score (GAD-7 scale)
  Interventions: Other: Attentional tasks

INTERVENTIONS:
Other: Attentional tasks — a neuropsychological assessment of attentional task, executive task and interview is proposed to patients or normal control

SUMMARY:
Epilepsy is one of the most common chronic neurological conditions.It leads to cognitive impairment in 20-50% of patients with a structural form.

In comparison with seizures, these cognitive disorders are a major additional factor in occupational, social and family disability. They are particularly frequent (50%) in temporal epilepsies and preferably concern memory and language skills.

The cognitive consequences of epilepsy are therefore well described in the following areas: episodic memory, language, executive functions.

Concerning attentional abilities, a recent review has highlighted the lack of work in this specific field in order to properly measure the prevalence and nature of attentional disorders in epileptic patients. Indeed, attentional abilities are often mentioned in studies, but attention is a complex domain defined by four modalities: alertness, selective attention, divided attention and sustained attention. No study systematically assesses all of these modalities.

The objective of this study is to evaluate the prevalence and nature of attentional disorders in epileptic patients compared to control subjects.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Patient with epilepsy, according to Fisher et al. (2005).
* Patient with written informed consent
* affiliation to a social security regime is compulsory
* Individuals who have received full information about the organization of the research and have not objected to their participation and the use of their data.
* Patient 18 years of age and older

Normal controls:

Individuals who have received full information about the organization of the research and have not objected to their participation and the use of their data.

* People 18 years of age and older
* People with no neurological and/or psychiatric history

Exclusion Criteria:

for patients: with another progressive neurological condition for all People of full age who are subject to a legal protection measure or who are unable to express their consent People deprived of their liberty by a judicial or administrative decision People who regularly use psychoactive substances (cannabis, alcohol...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with epilepsy versus normal control
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
d2-r | 10 minutes
  selective attention task

SECONDARY OUTCOMES:
sustained attention TAP Subtest | 15 minutes
  Your task is to press the key as quickly as possible whenever two successive patterns have the same shape
alertness attention TAP Subtest | 8 minutes
  a cross appears on the screen. press the key when the cross appears
divided attention TAP Subtest | 5 minutes
  first task :a cross appears on the screen in which a varying number of crosses appear simultaneously. when four of these crosses form a square, then please press the key as quickly as possible.
  second task: in this task you will hear a high and a low tone in sequence. you must decide whether the same tone occurs twice in a row. Please press the key as quickly as possible.

OTHER OUTCOMES:
digit span | 5 minutes
  immediate memory task
verbal fluency | 5 minutes
  executive task
incompatibility TAP subtest | 8 minutes
  executive task
flexibility TAP subtest | 8 minutes
  executive task
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) | 3 minutes
  Depression scale score 0 to 24
GENERALIZED ANXIETY DISORDER (GAD-7) | 3 minutes
  ANXIETY scale score : 0 to 21

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brissart H, Forthoffer N, Maillard L. Attention disorders in adults with epilepsy. Determinants and therapeutic strategies. Rev Neurol (Paris). 2019 Mar;175(3):135-140. doi: 10.1016/j.neurol.2019.01.394. Epub 2019 Feb 28. PMID 30826090

DOCUMENTS (1):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT04379128/Prot_000.pdf